CLINICAL TRIAL: NCT07285954
Title: A Randomized Controlled Trial of a Walking Meditation Intervention (iWalk) to Enhance Resilience in Adults
Brief Title: Mindfulness Walking Intervention to Enhance Resilience (iWalk)
Acronym: iWalk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Chung-Yi Chiu, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-0202
Record Dates: First submitted 2025-10-16; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Neurodegenerative Disease; EEG; Mindfulness; Adults
Keywords: Walking meditation; Emotional regulation; EEG
MeSH Terms: conditions — Neurodegenerative Diseases; Emotional Regulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iWalk Program (Active Comparator): This group receives the complete iWalk program.
  Interventions: Behavioral: iWalk Program
- Education Only without Walking Mindfulness Practice (Active Comparator): This group receives only education part of the iWalk program without walking mindfulness sessions.
  Interventions: Behavioral: iWalk Program
- Control Group (No Intervention): This group does not receive any intervention and are placed on a waiting list.

INTERVENTIONS:
Behavioral: iWalk Program — A multi-component behavioral program integrating walking meditation, education, and group sessions to enhance resilience and stress regulation in adults with and without chronic conditions.
  Arms: Education Only without Walking Mindfulness Practice; iWalk Program

SUMMARY:
This study is a randomized controlled trial of the walking meditation intervention (iWalk) program, a multi-component intervention integrating walking meditation, education, and group sessions designed to enhance resilience in individuals with multiple sclerosis (MS).

The objectives are to evaluate:

1. Recruitment capability and retention rates,
2. Acceptability and adherence to the intervention,
3. Feasibility of assessment procedures, and
4. Preliminary effects on psychological, physiological, and behavioral outcomes.

DETAILED DESCRIPTION:
The iWalk Program is an 8-week, multi-component behavioral intervention integrating mindfulness-based stress reduction and walking meditation to promote resilience and self-regulation in people with MS. The intervention combines weekly educational content, guided walking meditation, and group reflection delivered both in-person and virtually. Participants in the experimental group will attend three one-hour sessions per week (two via Zoom, one in-person) focusing on mindfulness, interoception, emotional regulation, and positive coping.

The waitlist control group will receive usual care during the trial period and will be offered participation after study completion.

Assessments include psychological questionnaires, electroencephalography (EEG), cognitive tasks, balance testing, and physical activity monitoring using Fitbit and Hexoskin wearable sensors. Data analysis includes assessing quantitative and qualitative changes in resilience, stress, mindfulness, mood, interoceptive awareness, quality of life, and physical activity over 8 weeks.

The total study duration is 10 weeks per participant, including baseline and post-intervention assessments.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older,
2. clinical diagnosis of a neurodegenerative disease such as multiple sclerosis, Alzheimer's disease, Parkinson's disease, stroke, etc.,
3. have not practiced meditation regularly (e.g., 10 mins per day) and have never attended any meditation classes or community programs,
4. never received meditation training via coaching/certification/life coaching,
5. have internet access,
6. with no severe cognitive impairment, i.e., have a score of ≥ 21 on Modified Telephonic Interview for Cognitive Status (TICS-M),
7. be able to walk with or without an assistive device (Patient determined Disease Steps score ranged from 0-6),
8. are willing to be randomized to an intervention or a control group,
9. are willing to wear Fitbit (a wrist smart watch) for eight weeks,
10. are individuals who are right-handed according to the Edinburgh Handedness Questionnaire,
11. are willing to participate in all assessments, including in-person testing using electroencephalography (EEG) and cognitive tests, online survey/questionnaires, and online interviews or focus group discussions,
12. are willing to wear a Hexoskin t-shirt, which is a heart rate variability monitor, while doing the assessments in person.

Exclusion Criteria:

Participants who cannot speak, read, write, or listen in English.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Connor Davidson Resilience Scale for Adults (CD-RISC 25) | The baseline means assessments done two weeks before the intervention start date. Post-intervention assessments will be conducted two weeks after the intervention. Follow-up 1 is 24 weeks from baseline, and follow-up 2 is 48 weeks from baseline.
Multiple Sclerosis Resilience Scale (MSRS) | The baseline means assessments done two weeks before the intervention start date. Post-intervention assessments will be conducted two weeks after the intervention. Follow-up 1 is 24 weeks from baseline, and follow-up 2 is 48 weeks from baseline.
Stroop Task | The baseline means assessments done two weeks before the intervention start date. Post-intervention assessments will be conducted two weeks after the intervention. Follow-up 1 is 24 weeks from baseline, and follow-up 2 is 48 weeks from baseline.
Symbol Digit Modalities Test | The baseline means assessments done two weeks before the intervention start date. Post-intervention assessments will be conducted two weeks after the intervention. Follow-up 1 is 24 weeks from baseline, and follow-up 2 is 48 weeks from baseline.
Wisconsin Card Sorting Test | The baseline means assessments done two weeks before the intervention start date. Post-intervention assessments will be conducted two weeks after the intervention. Follow-up 1 is 24 weeks from baseline, and follow-up 2 is 48 weeks from baseline.
Sustained Attention to Response Task | The baseline means assessments done two weeks before the intervention start date. Post-intervention assessments will be conducted two weeks after the intervention. Follow-up 1 is 24 weeks from baseline, and follow-up 2 is 48 weeks from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No